CLINICAL TRIAL: NCT05081128
Title: A Placebo-Controlled Efficacy in iNPH Shunting (PENS) Trial
Brief Title: Efficacy in iNPH Shunting (PENS) Trial
Acronym: PENS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00305245; 1U01NS122764 (NIH); PENS (Other: Johns Hopkins University Department of Neurosurgery)
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus (INPH)

STUDY DESIGN:
Intervention Model Description: The primary intervention will be the initiation of the randomized initial shunt valve opening pressure setting to create a delayed treatment group in half of the study patients.
  Randomization will be to active or placebo (closed) shunt settings. At the time of the standard three-month evaluation, all subjects will be similarly non-invasively adjusted to bring all subjects in both groups to the active setting while maintaining blinding of the subjects. All settings will be verified by the adjusting neurosurgeon.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Open Shunt Group (Active Comparator): FDA-approved Certas Plus with Siphonguard, programmable CSF shunt valve setting to active (open shunt group)(setting 4)(110 mm H2O) at time of shunt implantation
  Interventions: Device: programmable CSF shunt valve
- Closed Shunt Group (Sham Comparator): FDA-approved Certas Plus with Siphonguard, programmable CSF shunt valve setting to placebo (closed shunt group)(setting 8)(>400 mm H2O) at time of shunt implantation followed by setting to active (setting 4) (110 mm H2O) three months after the procedure.
  Interventions: Device: programmable CSF shunt valve

INTERVENTIONS:
Device: programmable CSF shunt valve — Brain shunt surgery using a programmable CSF shunt valve
  Other Names: FDA-approved Certas Plus with Siphonguard

SUMMARY:
The Placebo-Controlled Efficacy in Idiopathic Normal Pressure Hydrocephalus (iNPH) Shunting (PENS) trial is a multi-center blinded, randomized, placebo-controlled design investigation of cerebrospinal fluid (CSF) shunt surgery to study the shunt efficacy in iNPH patients.

DETAILED DESCRIPTION:
The primary intervention will be setting the FDA-approved Certas Plus with Siphonguard, programmable CSF shunt valve to active (open shunt group)(setting 4)(110 mm H2O) or placebo (closed shunt group)(setting 8)(>400 mm H2O)in a 1:1 ratio. By the time of the primary objective evaluation at three months, the closed shunt group will have zero months of active treatment, and the open shunt group will have three months of active treatment. At three months, shunts for subjects in the closed shunt group will be adjusted to setting 4. To maintain blinding, all patients will be adjusted / mock adjusted to the active setting in a similar fashion. Patients from both groups will not be adjusted before three months of active treatment, unless judged medically necessary by the treating team. Following the three month visit, all subjects in each group will have shunt adjustments according to clinical standards at each center.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years; and
2. Diagnosis of iNPH and recommendation for shunt surgery based on the Investigator's clinical judgement based on criteria and testing as described in the iNPH Guidelines;
3. Evans Ratio ≥ 0.30; and
4. One positive supplementary test to include either large volume Lumbar Puncture or extended CSF drainage per institutional standards; and
5. History or evidence of gait impairment (such as decreased step height or length, decreased speed, retropulsion as described in the iNPH Guidelines) duration ≥ 6 months; and
6. Participant has the sensory motor skills, communication skills and understanding to comply with the testing and reporting required in the PENS trial; and
7. Participant is able to give written informed consent.

Exclusion Criteria:

1. Unable to walk 10 meters with or without an assistive device; or
2. Baseline fastest gait velocity (out of three gait trials) >1 m/sec prior to drainage trial and fastest gait velocity improvement is < 30% with or without an assistive device; or
3. Unable to return to the study center for follow up evaluation and shunt programming; or
4. Participant is not medically cleared for shunt surgery per local standards; or
5. Secondary NPH. (Prior encephalitis, meningitis, subarachnoid hemorrhage, traumatic brain injury (including concussion) within two years or with brain injury or skull fracture on baseline imaging, brain abscess, brain tumor, obstructive hydrocephalus (including acquired aqueductal stenosis and carcinomatous meningitis); or
6. Prior or existing shunts, endoscopic third ventriculostomy, or any previous surgical intervention for hydrocephalus; or
7. Previous intracranial neurosurgical procedure; or
8. Symptomatic cerebral or cerebellar infarction occurring within 6 months from screening (asymptomatic lacunar infarctions are permitted); or
9. Diagnosis of Parkinsonian syndrome that, in the investigator's judgment, will complicate the outcome evaluation; or
10. Diagnosis of schizophrenia or any psychiatric diagnosis (including depression) that, in the investigator's judgment, will complicate the outcome evaluation (such as neuroleptic treatment for schizophrenia); or
11. Diagnosis of dementia disorder where the investigator considers cognition deficit limits participation in the study; or
12. Conditions impairing gait that are considered to be unrelated to hydrocephalus, such as hemiparesis, spasticity, cerebellar ataxia or musculoskeletal and joint disease, which will interfere with gait assessment or the potential for gait improvement.
13. Individuals with contraindication to MRI (e.g., implanted electric and electronic devices, aneurysm clip(s), any metallic fragment or foreign body, coronary and peripheral artery stents, cardiac pacemaker, known claustrophobia, or known/possible pregnancy or breast-feeding) will be excluded according to institutional guidelines.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Gait velocity | Baseline and 3 months
  Evaluation of CSF shunting in iNPH patients through a group comparison of change from baseline at three months between active and placebo-controlled groups, using the primary endpoint of gait velocity (in meters per second).

SECONDARY OUTCOMES:
Cognition as assessed by the Montreal Cognitive Assessment (MoCA) | Baseline and 3 months
  Evaluate the effect of shunting between active and placebo-controlled groups at three months using MoCA test to assess cognition. Scores on the MoCA range from 0 to 30, with a score of 26 and higher generally considered normal.
Bladder Control as assessed by the Overactive Bladder Questionnaire, short form | Baseline and 3 months
  Evaluate the effect of shunting between active and placebo-controlled groups at three months using Overactive Bladder Questionnaire, short form (OAB-q sf.) to assess bladder control. The OAB-q sf consists of three QOL domains: coping, sleep, and emotional/social interaction. All scale scores are transformed to a 0- to 100-point scale, with lower scores indicating greater effect, i.e., worse QOL.
Balance and Gait as assessed by the Tinetti Score | Baseline and 3 months
  Evaluate the effect of shunting between active and placebo-controlled groups at three months using Tinetti Score to assess balance and gait. Scores on the Tinetti range from 0 to 28. The higher the score the better the gait and balance performance.

OTHER OUTCOMES:
Bladder Control as assessed by the Overactive Bladder Questionnaire, short form | Baseline and 12 months of active shunting
  Evaluate the effect of shunting between active and placebo-controlled groups at nine months using Overactive Bladder Questionnaire, short form (OAB-q sf.) to assess bladder control. All scale scores are transformed to a 0- to 100-point scale, with lower scores indicating greater effect, i.e., worse QOL.
Change in Gait velocity | Baseline and 12 months of active shunting
  Evaluate the change in gait velocity among all study participants between baseline and 12 months of active shunting, using the primary outcome of gait velocity (in meters per second).
Cognition as assessed by the Montreal Cognitive Assessment (MoCA) | Baseline and 12 months of active shunting
  Evaluate the effect of shunting between active and placebo-controlled groups at nine months using MoCA test to assess cognition. Scores on the MoCA range from zero to 30, with a score of 26 and higher generally considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Luciano, MD, PhD, Principal Investigator — Johns Hopkins University; Richard Holubkov, PhD, Study Director — University of Utah
Locations (17):
- United States (14):
  - University of California, Davis, Davis, California
  - University of Southern California, Los Angeles, California
  - Pacific Neuroscience Institute, Santa Monica, California
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - New York University Langone Health, New York, New York
  - Mount Sinai Health System, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver
- Umeå University, Umeå, Sweden

REFERENCES:
- [Derived] Luciano MG, Williams MA, Hamilton MG, Katzen HL, Dasher NA, Moghekar A, Hua J, Malm J, Eklund A, Alpert Abel N, Raslan AM, Elder BD, Savage JJ, Barrow DL, Shahlaie K, Jensen H, Zwimpfer TJ, Wollett J, Hanley DF, Holubkov R; PENS Trial Investigators and the Adult Hydrocephalus Clinical Research Network. A Randomized Trial of Shunting for Idiopathic Normal-Pressure Hydrocephalus. N Engl J Med. 2025 Dec 4;393(22):2198-2209. doi: 10.1056/NEJMoa2503109. Epub 2025 Sep 16. PMID 40960253